CLINICAL TRIAL: NCT06949488
Title: Efficacy of Dexmedetomidine, Dexamethasone, and Magnesium Sulphate as Adjuvants in Ultrasound-guided Supraclavicular Brachial Plexus Block in Forearm Surgeries - A Randomized Clinical Trial
Brief Title: Efficacy of Different Medications as Adjuvants in Ultrasound-guided Supraclavicular Brachial Plexus Block in Forearm Surgeries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohammed Gaber Saad, Lecturer of anesthesia, Intensive care and pain management., Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RHDIRB2018122002
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Upper Limb Surgery; Brachial Plexus Blockade
Keywords: Brachial Plexus Blockade; Mangesuim sulphate; ultrasound; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (DT): Dexmedetomidine group (Experimental): A group of 35 participants will receive 18 ml of bupivacaine 0.5% plus dexmedetomidine 100 µg for the supraclavicular block.
  Interventions: Procedure: Group A (DT): Dexmedetomidine group
- Group B (MG): Magnesium group (Experimental): A group of 35 participants will receive 18 ml of bupivacaine 0.5% plus magnesium sulfate 150 mg in 2 ml of normal saline for the same block.
  Interventions: Procedure: Group B (MG): Magnesium group
- Group C (DM): Dexamethasone group (Active Comparator): A group of 35 participants will receive 18 ml of bupivacaine 0.5% plus dexamethasone 8 mg for the same block.
  Interventions: Procedure: Group C (DM): Dexamethasone group

INTERVENTIONS:
Procedure: Group A (DT): Dexmedetomidine group — The ultrasound probe is placed in the supraclavicular fossa in the transverse orientation parallel to the clavicle and aimed inferior toward the ipsilateral thorax. The brachial plexus and the subclavian artery are visualized. The first rib appears as a hyperechoic line with the lung pleura deeper to this bony border. Utilizing the in-plane approach, the needle is advanced from lateral to medial, aimed near the main neural cluster of the brachial plexus. After negative aspiration, local anesthetic, including 100 µg Dexmeditomidine and normal saline, with a total volume of 20 mL, is injected. Subsequently, smaller aliquots of local anesthetic are deposited near the surrounding satellite neural clusters.
  Arms: Group A (DT): Dexmedetomidine group
Procedure: Group B (MG): Magnesium group — The ultrasound probe is placed in the supraclavicular fossa in the transverse orientation parallel to the clavicle and aimed inferior toward the ipsilateral thorax. The brachial plexus and the subclavian artery are visualized. The first rib appears as a hyperechoic line with the lung pleura deeper to this bony border. Utilizing the in-plane approach, the needle is advanced from lateral to medial, aimed near the main neural cluster of the brachial plexus. After negative aspiration, local anesthetic, including 150 mg of magnesium sulfate and normal saline, with a total volume of 20 mL, is injected. Subsequently, smaller aliquots of local anesthetic are deposited near the surrounding satellite neural clusters.
  Arms: Group B (MG): Magnesium group
Procedure: Group C (DM): Dexamethasone group — The ultrasound probe is placed in the supraclavicular fossa in the transverse orientation parallel to the clavicle and aimed inferior toward the ipsilateral thorax. The brachial plexus and the subclavian artery are visualized. The first rib appears as a hyperechoic line with the lung pleura deeper to this bony border. Utilizing the in-plane approach, the needle is advanced from lateral to medial, aimed near the main neural cluster of the brachial plexus. After negative aspiration, local anesthetic, including 8 mg dexamethasone and normal saline, with a total volume of 20 mL, is injected. Subsequently, smaller aliquots of local anesthetic are deposited near the surrounding satellite neural clusters.
  Arms: Group C (DM): Dexamethasone group

SUMMARY:
This study is to evaluate whether addition of dexmedetomidine, dexamethasone and magnesium sulfate as adjuvants to bupivacaine in supraclavicular Brachial Plexus Blockade (BPB) for pain management assessed by VAS score.

DETAILED DESCRIPTION:
This is a randomized controlled study involving 105 participants divided into three groups to assess the efficacy of adding dexmedetomidine, dexamethasone, and magnesium sulfate as adjuvants to bupivacaine in supraclavicular brachial plexus blockade during upper limb surgeries. The primary outcome is the postoperative Visual Analog Scale (VAS) score. The secondary outcomes are assessment of onset and duration of the block, patient satisfaction, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status of I and II
* undergoing forearm surgeries

Exclusion Criteria:

* coagulopathies
* Local skin lesions
* Pregnancy
* Has a history of significant neurological, psychiatric, or neuromuscular disorders
* Patients refusing participation
* BMI > 40
* Patient with COPD. hypersensitivity or allergies to local anesthesia

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
-Post operative Visual analogue scale VAS score | Over 24 hours post operative starting from transeferring the patient to the recovery area.
  Assess post-operative VAS score at: T0 (after transferring to the recovery area), at T1: at two hours, T3: at four hours, T4: at six hours, T5: at eight hours, T6: at 10 hours, T7: at 12 hours, T8: at 16 hours, T9: at 20 hours, and T10 at 24 hours postoperatively.

SECONDARY OUTCOMES:
Onst of sensory block | Complete sensory block will be assessed every 5 min up to a maximum of 30 minutes
  Time in minutes from completing the block to complete sensory loss to sensation of a cold cotton pad relative to the contralateral limb.
Onset of motor block | Complete motor block will be assessed every 5 min up to a maximum of 30 minutes
  Time in minutes from completing the block up to the time when the patient is unable to overcome gravity relative to the contralateral arm.
Duration of the sensory block | Sensation will be assessed every 4 hours till return of normal sensation up to maximum 24 hours .
  Complete return of the sensation in the blocked limb relative to the contralateral arm.
duration of the motor block | Motor power will be assessed every 4 hours till return of normal sensation up to maximum 24 hourswill be assessed every 4 hours till return of normal sensation up to maximum 24 hours
  Complete return of the motor power in the blocked limb
Intraoperative mean arterial blood pressure | From positioning the patient to the block upto 90 minutes from removing the needle
  Mean arterial blood pressure in mmHg will be assessed at T0: baseline before patient positing for the block, at T1: just after removing the needle, at T2: at 30 minutes, T3: at 60 Minutes , and T4: at 90 minutes intraoperatively
Intraoperative Pulse rate. | From positioning the patient to the block upto 90 minutes from removing the needle
  pulse rate per minute will be assessed at T0: baseline before patient positing for the block, at T1: just after removing the needle, at T2: at 30 minutes, T3: at 60 Minutes, and T4: at 90 minutes intraoperatively
Post operative opioid consumption | Over 24 hours post operatively started form transferring the patient to the recovery area
  Postoperative total doses of pethidine in milligrams will be counted. For patients with a VAS score of more than 4, pethidine 50mg will be given intramuscularly.
Post operative Nausea and vomiting | Over 24 hours post operative starting from transferring to the recovery area.
  Nausea and vomiting attacks will be recorded over 24 hours postoperatively.
Postoperative transient neurologic symptoms | Over 48 hours post operative starting from transeferring to the recovery area.
  Dysesthesia will be assessed every 12 hours postoperatively and reported

CONTACTS AND LOCATIONS:
Overall Officials: Hend Mostafa Abosaifa, MD, Study Director — Al-Azhar University; Fatma Alzahraa Roshdy Elkemary, MD, Principal Investigator — Al-Azhar Unversity; Noha Mohamed Elsai, MD, Study Chair — Al-Azhar Unversity; Ain ELmarwa Abdelmonem Abdallah, MD, Principal Investigator — Al-Azhar Unversity; Nashwa Mohammed Ibrahiem, MD, Study Chair — Al-Azhar Unversity; Wafaa Abd Ali Elhadi, MD, Study Chair — Al-Azhar Unversity; Hanaa Said Rashed, MD, Principal Investigator — National liver institute Menofia University
Locations (1):
- Faculity of medicine - Al-Azhar University hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Begon S, Pickering G, Eschalier A, Dubray C. Magnesium increases morphine analgesic effect in different experimental models of pain. Anesthesiology. 2002 Mar;96(3):627-32. doi: 10.1097/00000542-200203000-00019. PMID 11873038
- [Background] Kara H, Sahin N, Ulusan V, Aydogdu T. Magnesium infusion reduces perioperative pain. Eur J Anaesthesiol. 2002 Jan;19(1):52-6. doi: 10.1017/s026502150200008x. PMID 11913804
- [Background] Herman J, Urits I, Eskander J, Kaye AD, Viswanath O. Correction: Adductor Canal Block Duration of Analgesia Successfully Prolonged With Perineural Dexmedetomidine and Dexamethasone in Addition to IPACK Block for Total Knee Arthroplasty. Cureus. 2020 Nov 16;12(11):c39. doi: 10.7759/cureus.c39. PMID 33209562
- [Background] Zoratto D, Phelan R, Hopman WM, Wood GCA, Shyam V, DuMerton D, Shelley J, McQuaide S, Kanee L, Ho AM, McMullen M, Armstrong M, Mizubuti GB. Adductor canal block with or without added magnesium sulfate following total knee arthroplasty: a multi-arm randomized controlled trial. Can J Anaesth. 2021 Jul;68(7):1028-1037. doi: 10.1007/s12630-021-01985-5. Epub 2021 May 26. PMID 34041719
- [Background] Bruce BG, Green A, Blaine TA, Wesner LV. Brachial plexus blocks for upper extremity orthopaedic surgery. J Am Acad Orthop Surg. 2012 Jan;20(1):38-47. doi: 10.5435/JAAOS-20-01-038. PMID 22207517